CLINICAL TRIAL: NCT05841992
Title: Comparison of the Detection Efficiencies of Al18F-PSMA-617 and 68Ga-PSMA-617 PET/CT in Patients With Prostate Cancer
Brief Title: Al18F-PSMA-617 and 68Ga-PSMA-617 PET/CT Imaging in the Same Group of Prostate Cancer Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCHFPSMA617
Record Dates: First submitted 2023-04-12; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Al18F-PSMA-617 and 68Ga-PSMA-617 PET/CTscan (Experimental): Patients of Prostate cancer PET/CT imaging: In two consecutive days each patient underwent a PET/CT scan after intravenous administration of 68Ga-PSMA617 and Al18F-PSMA-617, respectively.
  Interventions: Drug: Al18F-PSMA-617; Drug: 68Ga-PSMA-617

INTERVENTIONS:
Drug: Al18F-PSMA-617 — Intravenous injection of one dosage of 0.1mCi/kg Al18F-PSMA-617. Tracer doses of Al18F-PSMA-617 will be used to image lesions of prostate cancer by PET/CT.
  Other Names: Al18F-PSMA-617 injection
Drug: 68Ga-PSMA-617 — Intravenous injection of one dosage of 148-185 MBq (4-5 mCi) 68Ga-PSMA-617. Tracer doses of 68Ga-PSMA-617 will be used to image lesions of prostate cancer by PET/CT.
  Other Names: 68Ga-PSMA-617 injection

SUMMARY:
18F-labeled prostate-specific membrane antigen (PSMA) ligand-positron emission tomography (PET) offers advantages over 68Ga-labeled PSMA ligands. Al18F-PSMA-617 is a novel 18F-PSMA compound used for prostate cancer (PCa) imaging. This pilot study was prospectively designed to compare the lesion detectability of Al18F-PSMA-617 and related 68Ga-PSMA-617 PET/CT in patients with PCa

DETAILED DESCRIPTION:
Prostate cancer (PC) is one of the most common malignancies worldwide in men, with persistently high numbers dying from this disease. Due to low levels of glycolysis in prostate cancer cell, the uses of 18F-FDG PET/CT to detect prostate cancer and its metastases are limited. Prostate specific membrane antigen (PSMA), as known as folate hydrolase I or glutamate carboxypeptidase II, is overexpressed on the cells of prostatic adenocarcinoma. Various low molecular weight radiopharmaceuticals targeting PSMA such as PSMA-617, PSMA-11 for 68Ga-labeling have been developed. 68Ga-PSMA PET/CT has demonstrated desirable sensitivity and specificity in the detection of prostate cancer lesions, which can find many micro lesions that cannot be identified by CT, MRI and bone scan. Al18F-PSMA-617 is a novel radiopharmaceutical targeting PSMA. Liu T et.al had demonstrated that Al18F-PSMA-617 accumulates specifically in PSMA-positive tumors with high binding affinity and selectivity. The first in-human evaluation of Al18F-PSMA-617 in a small PCa sample size also confirmed the good detectability of tumor lesions. This pilot study was prospectively designed to evaluate the early dynamic distribution of Al18F-PSMA-617 compared with 68Ga-PSMA-617 in the same group of prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* confirmed untreated prostate cancer patients;

  * 68Ga-PSMA617 and Al18F-PSMA-617 PET/CT within two consecutive days;
  * signed written consent.

Exclusion Criteria:

* known allergy against PSMA; • any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Time-activity curves | through study completion, an average of 1 year
  During the early dynamic Al18F-PSMA-617 PET imaging, the SUVmax of PCa lesions, the SUVmean of the normal tissues such as the prostate gland , the common iliac artery , the bladder, and the gluteus maximus were measured.Time-activity curves(TACs) describing SUVmax versus time of tumor lesion and areas with physiologic tracer uptake were generated.
Kinetic parameters | through study completion, an average of 1 year
  Based on dynamic Al18F-PSMA-617 PET imaging, tracer kinetics(k1,k2,k3,k4,ki ) in tumor and normal tissues were generated by means of a two-tissue irreversible compartment model and Patlak graphical analysis.
Differences in lesion detection at different imaging time point | through study completion, an average of 1 year
  In addition to the early dynamic images, we also performed whole-body delayed imaging at 2h and 4h after injection of Al18F-PSMA-617.The differences in lesion detectability at different time point were compared in order to determine the optimal imaging time.
Diagnostic value | hrough study completion, an average of 1 year
  Sensitivity and Specificity of Al18F-PSMA-617 PET/CT for prostate cancer in comparison with 68Ga-PSMA-617

SECONDARY OUTCOMES:
SUVmax of tumor | through study completion, an average of 1 year
  The tumor uptake on Al18F-PSMA-617 PET/CT for prostate cancer in comparison with 68Ga-PSMA-617 PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Li Huo, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China